CLINICAL TRIAL: NCT04454632
Title: Examination of the Effectiveness of Mirror Therapy in the Treatment of Patients With Frozen Shoulder: A Prospective Randomized Controlled Study
Brief Title: The Effect of Mirror Therapy in Patients With Frozen Shoulder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Marmara University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: Dr. Lutfi Kirdar Hospital
Record Dates: First submitted 2020-06-25; First posted 2020-07-01 (Actual); Last update posted 2021-06-10 (Actual); Status verified 2020-06

CONDITIONS: Pain; Frozen Shoulder
Keywords: Frozen Shoulder; visual feedback; proprioception; pain insensitivity; shoulder pain
MeSH Terms: conditions — Pain; Bursitis; Agnosia; Shoulder Pain | interventions — Mirror Movement Therapy; Feedback, Sensory

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Mirror therapy group (Experimental): The number of participants in this group is anticipated to be 12. In addition to basic treatment, the mirror therapy group bilateral exercised with the affected arm behind the mirror for 10 minutes after every session. Participants in this group perform three exercises as glenohumeral flexion, abduction, and rotation.
  Interventions: Other: Mirror therapy
- Visual feedback group (Experimental): The number of participants in this group is anticipated to be 12. In addition to basic treatment, the visual feedback group bilateral exercised by seeing both arms in the mirror for 10 minutes after every session. Participants in this group perform three exercises as glenohumeral flexion, abduction, and rotation while seeing both arms in the mirror.
  Interventions: Other: Visual feedback
- Control group (No Intervention): The number of participants in this group is anticipated to be 12. In addition to basic treatment, the control group bilateral exercised without a mirror for 10 minutes after every session. Participants in this group perform three exercises as glenohumeral flexion, abduction, and rotation while seeing both arms in the mirror.

INTERVENTIONS:
Other: Mirror therapy — affected arm stay behind the mirror while exercising
  Arms: Mirror therapy group
Other: Visual feedback — visual feedback from mirror
  Arms: Visual feedback group

SUMMARY:
The aim of this study compares mirror therapy and visual feedback treatment with the control group in frozen shoulder patients.

DETAILED DESCRIPTION:
Thirty-six individuals divided three groups as mirror therapy, visual feedback, and control groups were included in the study for 15 sessions of treatment. All individuals received basic treatment as ultrasound, transcutaneous electrical nerve stimulation, cold pack, stretching exercises, glenohumeral range of motion exercises, scapulothoracic exercises. The mirror group bilateral exercised with an affected arm behind the mirror; visual feedback group bilateral exercised by seeing both arms in the mirror; control group bilateral exercised without a mirror for 10 minutes after every session. Pain severity was evaluated with the "Visual Analogue Scale (VAS)", ROM and proprioception were measured with a universal goniometer, and functional status was evaluated with "shoulder pain and disability index (SPADI)" and "Modified Constant Score". Evaluations were made before, day after the treatment and 4 weeks after the treatment by the same researcher. Data analysis was performed with SPSS.23.

ELIGIBILITY:
Inclusion Criteria:

* Individuals who were diagnosed with "Unilateral Frozen Shoulder" by the specialist;
* Normal radiological imaging;
* Aged between 18-75 years old;
* Symptoms persist for 2-12 months.

Exclusion Criteria:

* If patients had following comorbidities: rotator cuff injury, cervical radiculopathy, romatological diseases, neurological diseases, fracture, tumour, congenital deformities, dislocation or sublocation, surgery in the shoulder, uncontrolled hypertension or diabetes mellitus;
* Pregnancy;
* Patients who had previously received physical therapy;
* Patients having problems in the perception of tests and exercises were excluded from this study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2018-02-15 (Actual); Primary Completion 2019-05-29 (Actual); Study Completion 2019-06-27 (Actual)

PRIMARY OUTCOMES:
Visual Analog Scale (VAS) | Change from Baseline, 6 weeks and 10 weeks
  Pain intensity was obtained using a Visual Analog Scale (VAS). VAS is usually a horizontal line, 10 cm in length, anchored by word descriptors at each end with "No Pain" (score of zero) on the left side up to "severe pain" on the right side. The patient was asked to mark the line point that represented his or her worst pain in the past week during daily rutine.
Range of Motion (ROM) | Change from Baseline, 6 weeks and 10 weeks
  Range of motion is the measurement of the amount of movement around a joint as a flexion, abduction, external rotation and internal rotation (degree). Measurement performed with universal goniometer.
Proprioception | Change from Baseline, 6 weeks and 10 weeks
  Proprioception is the sense of self-movement and body position. A joint position error test (JPET) was used for proprioception measurement. JPET is a deviation of the ability to reposition the joint to the target position which fifty percent of active flexion ROM.
Shoulder Pain and Disability Index (SPADI) | Change from Baseline, 6 weeks and 10 weeks
  The shoulder pain and disability index is a self-administered questionnaire that consists of two dimensions, one for pain and the other one for functional activities on the shoulder. The total score is defining as a percent. 0 for best score 100 for worst score.
Modified Constant-Murley Score (CMS) | Change from Baseline, 6 weeks and 10 weeks
  The modified Constant-Murley score is a questionnaire for shoulder injuries that consists of four dimensions, pain, activities of daily living, range of movement, and power. Pain and activities of daily living are considered subjective scores therefore the range of movement and power considered objective score. 100 for best score 0 for worst score.

CONTACTS AND LOCATIONS:
Overall Officials: TUGBA KURU ÇOLAK, Assoc. Prof., Study Director — Marmara University
Locations (1):
- Dr. Lutfi Kirdar City Hospital, Istanbul, Kartal, Turkey (Türkiye)

REFERENCES:
- [Result] Baskaya MC, Ercalik C, Karatas Kir O, Ercalik T, Tuncer T. The efficacy of mirror therapy in patients with adhesive capsulitis: A randomized, prospective, controlled study. J Back Musculoskelet Rehabil. 2018;31(6):1177-1182. doi: 10.3233/BMR-171050. PMID 30056414
- [Result] Sato K, Fukumori S, Matsusaki T, Maruo T, Ishikawa S, Nishie H, Takata K, Mizuhara H, Mizobuchi S, Nakatsuka H, Matsumi M, Gofuku A, Yokoyama M, Morita K. Nonimmersive virtual reality mirror visual feedback therapy and its application for the treatment of complex regional pain syndrome: an open-label pilot study. Pain Med. 2010 Apr;11(4):622-9. doi: 10.1111/j.1526-4637.2010.00819.x. Epub 2010 Mar 1. PMID 20202141
- See also: Mirror therapy in frozen shoulder — https://pubmed.ncbi.nlm.nih.gov/30056414/
- See also: visual feedback therapy — https://pubmed.ncbi.nlm.nih.gov/20202141/